CLINICAL TRIAL: NCT06817057
Title: The Effect of Virtual Reality on the Patient Experience During Wide-Awake Hand Surgery: A Randomised Controlled Trial
Brief Title: Virtual Reality in Wide-Awake Hand Surgery
Acronym: VR-WAHS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Researchers left institution
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 292555
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Virtual Reality; Upper Extremity Problem
Keywords: Virtual Reality; VR; Wide-Awake Hand Surgery; WAHS; Upper Extremity; Upper Limb; Local Anaesthesia; Regional Anaesthesia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WITH Virtual Reality headset + headphones (Experimental): Participants in the VR arm will undergo wide-awake hand surgery while using an Oculus Quest 2 Virtual Reality headset and Beats Ep Wired On-Ear headphones for the duration of the operation, as an adjunct to standard local or regional anaesthesia.
  Interventions: Device: Virtual Reality headset + headphones
- WITHOUT Virtual Reality headset + headphones (No Intervention): Participants in the non-VR arm will undergo wide-awake hand surgery under the conditions of routine intraoperative care, that is under local or regional anaesthesia without any adjuncts, such as the Virtual Reality headset, headphones, or any other form of distraction or relaxation strategy.

INTERVENTIONS:
Device: Virtual Reality headset + headphones — The intervention involves patient use of a Virtual Reality headset (the Oculus Quest 2) and headphones (Beats Ep Wired On-Ear) during their wide-awake hand operation.
  Other Names: Oculus Quest 2 Virtual Reality Headset + Beats Ep Wired On-Ear Headphones
  Arms: WITH Virtual Reality headset + headphones

SUMMARY:
The vast majority of hand surgery performed at the Royal London Hospital is carried out with patients wide-awake. This is either using local or regional (brachial block) anaesthesia. A high proportion of patients find the process stressful and intimidating, which can lead to intraoperative anxiety and increased requirements for anaesthetic dosages. Most of the hand surgery lists are primarily performed by trainees under consultant supervision: conscious, aware, and anxious patients can hinder the degree of training that can take place intra-operatively. Trainees requesting for assistance can further contribute to patient anxiety levels. Virtual Reality (VR) is a relatively new technology that allows total immersion in audio-visual entertainment. Early research work has demonstrated a positive effect of VR at reducing patient anxiety and analgesia requirements during invasive procedures. The investigators hope to conduct a research study whereby adult patients undergoing wide-awake hand surgery under the care of the Department of Plastic Surgery at the Royal London Hospital are given a VR headset (the Oculus Quest 2) and headphones to wear during their operation. The investigators aim to compare their levels of perceived pain, discomfort, anxiety, relaxation and satisfaction with the intraoperative experience to patients who undergo the same operation without VR, i.e. under the conditions of standard care. The investigators will also look at the patients' additional anaesthetic requirements during the operation and physiological markers of anxiety, like heart rate and blood pressure. The operating surgeon will be given the opportunity to answer questions regarding their levels of comfort performing the operation, communicating with their assistant surgeon and calling for help if required. The investigators believe the use of VR will have a positive effect on the patient experience and will improve training opportunities for junior surgeons.

ELIGIBILITY:
Inclusion Criteria:

1. Written, informed consent provided prior to the occurrence of any study procedures;
2. Aged 18 years or above;
3. Undergoing a planned day-case operation involving the upper limb for any indication, under either local or regional anaesthesia.

Exclusion Criteria:

1. Suffer from claustrophobia, seizures or vertigo;
2. Have an active infection or open wound on the face;
3. Require droplet or airborne infection precautions;
4. Have eyesight or hearing problems that would impair the audio-visual experience of using VR (e.g. if the patient plans to wear hearing aids or eyeglasses during the operation);
5. Have a pacemaker or any other implanted medical device;
6. Are allergic to any materials on the VR headset or headphones (e.g. the VR headset facial interface foam).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Patient-reported Pain Score | Intraoperative score measured in the immediate postoperative period (<1 day)
  This will be measured by asking participants to rate their level of intraoperative pain along a 100-mm long visual analogue scale (0 - 100).
Patient-reported Discomfort Score | Intraoperative score measured in the immediate postoperative period (<1 day)
  This will be measured by asking participants to rate their level of intraoperative discomfort along a 100-mm long visual analogue scale.
Patient-reported Anxiety Score | Intraoperative score measured in the immediate postoperative period (<1 day)
  This will be measured by asking participants to rate their level of intraoperative anxiety along a 100-mm long visual analogue scale.
Patient-reported Relaxation Score | Intraoperative score measured in the immediate postoperative period (<1 day)
  This will be measured by asking participants to rate their level of intraoperative relaxation along a 100-mm long visual analogue scale.
Patient-reported Satisfaction Score | Intraoperative score measured in the immediate postoperative period (<1 day)
  This will be measured by asking participants to rate their level of overall satisfaction with their intraoperative experience along a 100-mm long visual analogue scale.

SECONDARY OUTCOMES:
Intraoperative Heart Rate | Intraoperative (<1 day)
  Mid-procedure heart rate measured in beats per minute
Intraoperative Blood Pressure | Intraoperative (<1 day)
  Mid-procedure systolic and diastolic blood pressure measured in millimetres of mercury
Additional Intraoperative Anaesthetic Doses | Intraoperative (<1 day)
  The type, dose and concentration of any additional doses of local anaesthesia given to the patient intraoperatively
Additional Intraoperative Sedative Doses | Intraoperative (<1 day)
  The type, dose and concentration of any (additional) doses of sedative medication given to the patient intraoperatively
Surgeon-reported Level of Comfort Performing the Operation | Intraoperative score measured in the immediate postoperative period (<1 day)
  This will be measured by asking the operating surgeon to rate their level of comfort performing the operation along a 100-mm long visual analogue scale.
Surgeon-reported Level of Comfort Communicating with Assistant Surgeon | Intraoperative score measured in the immediate postoperative period (<1 day)
  This will be measured by asking the operating surgeon to rate their level of comfort communicating with their assistant surgeon along a 100-mm long visual analogue scale.
Surgeon-reported Level of Comfort Calling for Help | Intraoperative score measured in the immediate postoperative period (<1 day)
  This will be measured by asking the operating surgeon to rate their level of comfort calling for help from a more senior surgeon along a 100-mm long visual analogue scale.

IPD SHARING:
Plan to Share IPD: No
No identifiable personal patient data will be shared with other researchers.